CLINICAL TRIAL: NCT06946537
Title: The Influence of Nutritional Status and Phenotypic Characteristics Upon Length of Stay, Clinical Outcome, and Survival in Hospitalized Patients
Brief Title: Nutritional Status and Patient Characteristics Upon Length of Stay, Clinical Outcome, and Survival in Older Hospitalized Patients
Acronym: INSIGHT
Status: Recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, Bispebjerg Hospital
Other Study IDs: H-25009586
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Geriatric; Malnutrition; Length of Stay
Keywords: Geriatric; Disease-related malnutrition; Physiology; Acute illness; Deep phenotyping; Nutritional status
MeSH Terms: conditions — Malnutrition | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (plasma and serum) and feces (fecal swabs)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The INSIGHT cohort: A geriatric cohort (age ≥ 65) established to investigate the coupling of phenotypical characteristics to nutritional and physiological status. The study intent to explore whether Disease-Related Malnutrition provides predictive value for patient prognosis based on specific phenotypic characteristics and establish different physiological stratifications to improve the identification of acutely admitted patients.
  Interventions: Other: Exposures and measurements

INTERVENTIONS:
Other: Exposures and measurements — Anthropometry, Body composition (BIA), Nutritional screening (GLIM, SNAQ, NIS, NRS-2002), Functional tests, Seisomocardiography, Muscle strength, Blood tests, Fecal swabs, Indirect calorimetry Orientation-Memory-Concentration (OMC), Sarcopenia, Frailty (Clinical Frailty Scale), Comobidity, Polypharmacy, Portrait photo.

SUMMARY:
Disease-related malnutrition (DRM) describes undernutrition or imbalances in energy, protein, or other nutrient-needs, caused by a concomitant disease. Nutritional status plays a vital role in the fate of hospitalized patients, and DRM is associated with loss of function and decreased survival.

DRM is a common condition in patients with acute illnesses, approximately 30% among medical inpatients are malnourished when admitteed to the hospital, and rise higher among the older or critically ill. Physiologically malnutrition is associated with a) poorer tissue healing and restitution after severe disease, b) suppressed immune function and resistance towards infections, c) poorer metabolic defense towards critical disease, d) delayed and poorer progress of chronic diseases. In addition, inadequate nutrition is coupled to a prolonged hospital stay, resulting in more readmissions, and overall higher mortality in hospital patients. Yet, nutritional status of patients upon hospital admittance is seldom systematically assessed and the consequences of DRM in older acutely admitted patients still needs to be understood.

This project will provide a detailed description of nutritional, physiolgical, and biochemical status of 1500 acutely admitted patients. In relation, the study will investigate the relation between patient characteristics and disease progression. The obtained data will also be coupled to patient registers to investigate the link between length of hospital stay, readmissions and acute contact, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted adults aged 65 years and above.
* Be able to comply with the study information, as assessed by the research personnel.
* Be able to understand Danish.

Exclusion Criteria:

* <24 hours admission
* Terminal illness in end stage of life
* Patients with temporary civil person registration number (CPR)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients acutely admitted at Bispebjerg Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay | From date of hospital admission untill discharge, assessed up to 2 months
  Time (in hours) hospitalized from arrival to discharge

SECONDARY OUTCOMES:
Readmission | Time to readmission 30 days from discharge
  Time to readmission from discharge
Acute contact | Time to acute contact 30 days from discharge
  Time to acute contact from discharge
Mortality | Time to mortality 90 days from index admission
  Time to mortality from index admission

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The following will be available: Study Protocol and Statistical Analysis Plan (SAP).